CLINICAL TRIAL: NCT01233102
Title: Umbilical Cord Mesenchymal Stem Cell Transfusion in Patients With Severe Liver Cirrhosis
Brief Title: Mesenchymal Stem Cells Treat Liver Cirrhosis
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yufang Shi (Other Government)
Collaborators: Soochow University (Other)
Responsible Party: Sponsor-Investigator, Yufang Shi, principal investigator, Chinese Academy of Sciences
Organization: Chinese Academy of Sciences (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIBS-IHS-20101010; 2010CB945600 (Other Grant/Funding Number: 2010CB945600-Chinese Ministry of Health)
Record Dates: First submitted 2010-10-25; First posted 2010-11-03 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Liver Cirrhosis
Keywords: liver Cirrhosis; Mesenchymal stem cells; Hepatic artery infusion; Intravenous infusion
MeSH Terms: conditions — Liver Cirrhosis | interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conserved Therapy (Active Comparator): Conserved Therapy
  Interventions: Drug: Conserved Therapy
- Interventional Therapy (Experimental): Patients with liver cirrhosis will be randomly divided into three groups.
  1. Umbilical cord MSCs will be infused to patients using interventional method via hepatic artery for one group.2. Umbilical cord MSCs will be infused to patients intravenously for another group. The control group will receive conserved therapy. The efficacy of different interventional therapies will be compared.
  Interventions: Procedure: Hepatic artery infusion or Intravenous infusion

INTERVENTIONS:
Drug: Conserved Therapy — Conserved Therapy
  Arms: Conserved Therapy
Procedure: Hepatic artery infusion or Intravenous infusion — Patients with liver cirrhosis will be randomly divided into three groups. Umbilical cord MSCs will be infused to patients using interventional method via hepatic artery for one group. The catheter will be inserted to proper hepatic artery. After the catheter placement confirmed by angiography, umbilical cord MSCs will be infused slowly in 20-30 minutes. Umbilical cord MSCs will be infused intravenously slowly for 30-60 minutes in the intravenous infusion group. The control group will receive conserved therapy.
  Arms: Interventional Therapy

SUMMARY:
The purpose of this study is to investigate the efficacy of umbilical cord mesenchymal stem cells (MSCs) transfusion in the treatment of liver cirrhosis. Liver function will be monitored by serum analysis. The levels of serum alanine aminotransferase (ALT), total bilirubin (TB), prothrombin time (PT), prealbumin(PA) and albumin (ALB) will be examined at pre-transfusion, and 3 days to 2 years post-transfusion. Child-Pugh scores, Model for End-Stage Liver Disease scores and clinical symptoms will be assessed simultaneously.

DETAILED DESCRIPTION:
Patients with liver cirrhosis will be randomly divided into three groups. Umbilical cord MSCs will be infused to patients using interventional method via hepatic artery for one group. The catheter will be inserted to proper hepatic artery. After the catheter placement confirmed by angiography, umbilical cord MSCs will be infused slowly in 20-30 minutes. Umbilical cord MSCs will be infused intravenously slowly in 30-60 minutes in the intravenous infusion group. The control group will receive conserved therapy. The levels of serum alanine aminotransferase (ALT), total bilirubin (TB), prothrombin time (PT), prealbumin(PA)and albumin (ALB) will be examined at re-transplantation, and 3 days to 2 years post-transplantation. The efficacy of umbilical cord MSCs transfusion will be investigated. The efficacy of different interventional therapies will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years.
* Imaging evidences of liver cirrhosis.
* Child-Plough score of 8 or more.
* Model for End-Stage Liver Disease score of 20 or more.

Exclusion Criteria:

* Liver tumor on ultrasonography, CT or MRI examination.
* Problems in organs other than liver (e.g. heart or lungs).
* History of moderate to severe hepatic encephalopathy or variceal bleeding.
* Imaging evidences of vascular thromboses.
* Coma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-10; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The level of serum alanine aminotransferase (ALT） | 1 year
The level of serum total bilirubin (TB) | 1 year
The level of serum prothrombin time (PT) | 1 year
The level of serum prealbumin(PA) | 1 year
The level of serum albumin (ALB) | 1 year
Overall survival | 1 year

SECONDARY OUTCOMES:
liver biopsy | 2 years
Overall survival | 2 years
The level of serum alanine aminotransferase (ALT） | 2 years
The level of serum total bilirubin (TB) | 2 years
The level of serum prothrombin time (PT) | 2 years
The level of serum albumin (ALB) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yufang Shi, PhD,DVM, Principal Investigator — Chinese Academy of Sciences; Jianhe Gan, MD, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

REFERENCES:
- [Background] Ren G, Zhang L, Zhao X, Xu G, Zhang Y, Roberts AI, Zhao RC, Shi Y. Mesenchymal stem cell-mediated immunosuppression occurs via concerted action of chemokines and nitric oxide. Cell Stem Cell. 2008 Feb 7;2(2):141-50. doi: 10.1016/j.stem.2007.11.014. PMID 18371435
- [Background] Terai S, Ishikawa T, Omori K, Aoyama K, Marumoto Y, Urata Y, Yokoyama Y, Uchida K, Yamasaki T, Fujii Y, Okita K, Sakaida I. Improved liver function in patients with liver cirrhosis after autologous bone marrow cell infusion therapy. Stem Cells. 2006 Oct;24(10):2292-8. doi: 10.1634/stemcells.2005-0542. Epub 2006 Jun 15. PMID 16778155
- [Background] Kharaziha P, Hellstrom PM, Noorinayer B, Farzaneh F, Aghajani K, Jafari F, Telkabadi M, Atashi A, Honardoost M, Zali MR, Soleimani M. Improvement of liver function in liver cirrhosis patients after autologous mesenchymal stem cell injection: a phase I-II clinical trial. Eur J Gastroenterol Hepatol. 2009 Oct;21(10):1199-205. doi: 10.1097/MEG.0b013e32832a1f6c. PMID 19455046
- [Background] Dai LJ, Li HY, Guan LX, Ritchie G, Zhou JX. The therapeutic potential of bone marrow-derived mesenchymal stem cells on hepatic cirrhosis. Stem Cell Res. 2009 Jan;2(1):16-25. doi: 10.1016/j.scr.2008.07.005. Epub 2008 Aug 6. PMID 19383405
- [Background] Abdel Aziz MT, Atta HM, Mahfouz S, Fouad HH, Roshdy NK, Ahmed HH, Rashed LA, Sabry D, Hassouna AA, Hasan NM. Therapeutic potential of bone marrow-derived mesenchymal stem cells on experimental liver fibrosis. Clin Biochem. 2007 Aug;40(12):893-9. doi: 10.1016/j.clinbiochem.2007.04.017. Epub 2007 May 3. PMID 17543295
- [Background] Li C, Kong Y, Wang H, Wang S, Yu H, Liu X, Yang L, Jiang X, Li L, Li L. Homing of bone marrow mesenchymal stem cells mediated by sphingosine 1-phosphate contributes to liver fibrosis. J Hepatol. 2009 Jun;50(6):1174-83. doi: 10.1016/j.jhep.2009.01.028. Epub 2009 Mar 29. PMID 19398237
- [Background] Kim TH, Kim JK, Shim W, Kim SY, Park TJ, Jung JY. Tracking of transplanted mesenchymal stem cells labeled with fluorescent magnetic nanoparticle in liver cirrhosis rat model with 3-T MRI. Magn Reson Imaging. 2010 Sep;28(7):1004-13. doi: 10.1016/j.mri.2010.03.047. PMID 20663626
- [Background] Rabani V, Shahsavani M, Gharavi M, Piryaei A, Azhdari Z, Baharvand H. Mesenchymal stem cell infusion therapy in a carbon tetrachloride-induced liver fibrosis model affects matrix metalloproteinase expression. Cell Biol Int. 2010 Apr 27;34(6):601-5. doi: 10.1042/CBI20090386. PMID 20178458